CLINICAL TRIAL: NCT07006610
Title: Comparison of the Effects of Hilotherapy and Kinesio Taping on Edema, Pain, and Trismus After Orthognathic Surgery
Brief Title: Hilotherapy vs. Kinesio Taping in Orthognathic Surgery Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ozge Sen, PhD Student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEDIPOL-BAP-2024-39; BAP-2024-39 (Other Grant/Funding Number: Istanbul Medipol University Scientific Research Projects Commission (BAP))
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Edema; Postoperative Pain; Trismus; Orthognathic Surgery
Keywords: Hilotherapy; Kinesio Taping; Orthognathic Surgery; Postoperative Complications; Postoperative Recovery
MeSH Terms: conditions — Pain, Postoperative; Trismus; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hilotherapy Group (Experimental): Participants in this group will receive hilotherapy applied one hour after orthognathic surgery. A polyurethane facial mask (Hilotherm® device) delivering continuously cooled water at +17°C will be worn for at least 16 hours per day, for a total of 48 hours. The therapy aims to reduce postoperative pain, edema, and trismus through controlled cooling.
  Interventions: Device: Hilotherm® Facial Cooling System
- Kinesio Taping Group (Experimental): Participants in this group will receive kinesio taping applied one hour after orthognathic surgery. The tapes (Kinesio Tex® Gold) will remain in place for 5 days (120 hours) without removal. The taping is intended to promote lymphatic drainage, reduce facial swelling, and improve functional recovery.
  Interventions: Device: Kinesio Tex® Gold Taping

INTERVENTIONS:
Device: Kinesio Tex® Gold Taping — Elastic kinesio tape applied postoperatively to the facial region and left in place for 5 days.
  Arms: Kinesio Taping Group
Device: Hilotherm® Facial Cooling System — A polyurethane facial mask delivering continuous +17°C water cooling for 48 hours post-surgery.
  Arms: Hilotherapy Group

SUMMARY:
This prospective randomized controlled trial aims to compare the effects of kinesio taping and hilotherapy on postoperative edema, pain, and trismus in patients undergoing bimaxillary orthognathic surgery.

DETAILED DESCRIPTION:
Orthognathic surgery frequently causes postoperative edema, pain, and trismus. The study compares two adjunctive therapies: kinesio taping and hilotherapy. Forty-four patients without systemic disease, undergoing Le Fort I + BSSRO, will be randomly assigned to two groups. Group 1 will receive kinesio taping for 5 days. Group 2 will undergo hilotherapy for 48 hours. Pain (VAS), trismus (mouth opening), and edema (measured by both tape and 3D scanner) will be assessed at multiple postoperative time points. The goal is to determine the more effective intervention for postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo bimaxillary orthognathic surgery (Le Fort I + BSSRO)
* Age between 18 and 50 years
* No systemic disease
* Voluntary participation with signed informed consent

Exclusion Criteria:

* Presence of systemic disease or immunosuppressive medication
* Known allergy to kinesio tape
* Inability to attend follow-up appointments
* Facial anatomical deformities preventing measurement

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Facial Edema | Baseline (Post-op 1.hour) and Post-op Days 1, 2, 5, 10, and 30
  Facial edema will be measured using both linear tape-based anthropometric measurements and 3D facial scanning at specified time points. Measurements will include tragus-to-ala, tragus-to-pogonion, and other standard facial distances.

SECONDARY OUTCOMES:
Change in Pain Score (VAS) | Baseline(Post-op 1.hour) and Post-op Days 1, 2, 5, 10, and 30 |
  Pain will be assessed using a 10-point Visual Analog Scale (VAS), with 0 indicating no pain and 10 indicating the worst imaginable pain.
Change in Trismus (Maximum Mouth Opening) | Baseline(Post-op 1.hour) and Post-op Days 1, 2, 5, 10, and 30
  Trismus will be assessed by measuring maximum interincisal distance using a millimeter ruler.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Mega Hospital, Istanbul, Bağcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is a single-center academic thesis project with a limited sample size and no data-sharing agreement is planned.

REFERENCES:
- [Background] Rana M, Gellrich NC, Joos U, Piffko J, Kater W. 3D evaluation of postoperative swelling using two different cooling methods following orthognathic surgery: a randomised observer blind prospective pilot study. Int J Oral Maxillofac Surg. 2011 Jul;40(7):690-6. doi: 10.1016/j.ijom.2011.02.015. Epub 2011 Mar 15. PMID 21411291
- [Background] Tozzi U, Santagata M, Sellitto A, Tartaro GP. Influence of Kinesiologic Tape on Post-operative Swelling After Orthognathic Surgery. J Maxillofac Oral Surg. 2016 Mar;15(1):52-8. doi: 10.1007/s12663-015-0787-0. Epub 2015 Mar 29. PMID 26929553
- [Background] Apostolov R, Asadi K, Lokan J, Kam N, Testro A. Mycophenolate mofetil toxicity mimicking acute cellular rejection in a small intestinal transplant. World J Transplant. 2017 Feb 24;7(1):98-102. doi: 10.5500/wjt.v7.i1.98. PMID 28280702
- [Background] Wei W, Zhao H, Wang A, Sui M, Liang K, Deng H, Ma Y, Zhang Y, Zhang H, Guan Y. A clinical study on the short-term effect of berberine in comparison to metformin on the metabolic characteristics of women with polycystic ovary syndrome. Eur J Endocrinol. 2012 Jan;166(1):99-105. doi: 10.1530/EJE-11-0616. Epub 2011 Oct 21. PMID 22019891
- [Background] Golkar M, Taheri A, Alam M, Asadi Y, Keyhan SO. The effects of Kinesio tapes on facial swelling following bimaxillary orthognathic surgery in the supraclavicular region. Maxillofac Plast Reconstr Surg. 2023 Jun 19;45(1):22. doi: 10.1186/s40902-023-00385-7. PMID 37335425